CLINICAL TRIAL: NCT03667469
Title: A Study of Life Expectancy in Patients With Metabolic Syndrome After Weight Loss: a Comparative Randomized Clinical Trial
Brief Title: Study of the Life Expectancy of Patients With Metabolic Syndrome After Weight Loss:
Acronym: LIFEXPE-RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center, Kazakhstan (Other)
Responsible Party: Principal Investigator, Oral Ospanov, Professor, University Medical Center, Kazakhstan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMC
Record Dates: First submitted 2018-08-31; First posted 2018-09-12 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Ospanov's procedure; One anastomosis gastric bypass; Stapleless - separated gastric bypass; Weight loss therapy; Metabolic syndrome; Life expectancy; Telomere lenght; Hypocaloric diet
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated to one of three groups:
  1. Surgical bariatric procedure in the first (A) group undergo the laparoscopic stapleless-separated mini-gastric bypass procedure: Gastric band (absorbable ligature) was introduced in the abdomen and retracted through the retrogastric tunnel. Mobilization and displacement of gastric fundus and create obstructive gastroplication. Hand-sewn gastrojejunostomy completes the intervention.
  2. Surgical bariatric procedure in the second (B) group: Linear cutter stapler-separated mini-gastric bypass (MGB/OAGB): standard surgery.
  3. Non-Surgical interventional in three (C) group including hypocaloric diet therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: sealed non-transparent envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stapleless one anastomosis gastric bypass (Experimental): Laparoscopic stapleless-separated one anastomosis (mini-) gastric bypass procedures
  Interventions: Procedure: Laparoscopic one anastomosis gastric bypass
- Staple use mini-gastric bypass (Active Comparator): Laparoscopic stapler-separated one anastomosis (mini-) gastric bypass procedures
  Interventions: Procedure: Laparoscopic one anastomosis gastric bypass
- Hypocaloric diet therapy (Active Comparator): Hypocaloric diet therapy with energy restriction (-500 kcal/d)
  Interventions: Dietary Supplement: Hypocaloric diet therapy

INTERVENTIONS:
Procedure: Laparoscopic one anastomosis gastric bypass — Laparoscopic surgical bariatric procedure with creation gastric pouch. A jejunal loop was created about 200 cm from the ligament of Treitz and anastomosed to the gastric pouch.
  Other Names: MGB/OAGB; mini-gastric bypass
  Arms: Staple use mini-gastric bypass; Stapleless one anastomosis gastric bypass
Dietary Supplement: Hypocaloric diet therapy — Hypocaloric diet therapy with energy restriction (-500 kcal/d)
  Arms: Hypocaloric diet therapy

SUMMARY:
Background and study aims:

Surgical and non-surgical normalization of body weight with obesity leads to a significant improvement in health and regression of metabolic syndrome. But as the reduction in body weight with obesity changes the life expectancy remains not clear enough.

The use of endoscopic staplers does not exclude the emergence of serious complications of surgery, for example, including bleeding and leakage in the stapler suture line. Therefore, the advantages of using a band in the bariatrics are justified from a security standpoint.

Currently, the gastric bypass is increasingly performed in the version of the mini gastric bypass (MGB). Another name for the procedure: one anastomosis gastric bypass (OAGB). The proposal to use for the staple-free (stepleless or steplerless) creation of a pouch (band-separated gastric bypass) with use for band a vascular prosthesis is justified, but it requires comparison of this method with a stapler variant.

An important issue is comparing surgical and non-surgical weight loss with obesity and metabolic syndrome and comparing life expectancy with confirmation of changes in telomere length.

This study compares loss of weight, changes in other health conditions that the patient may have (co-morbidities, such as diabetes), telomere length, quality of life, the number of complications and side effects, the degree of complexity of the surgical technique and operating costs of a new laparoscopic band-separated mini- gastric bypass (LBSMGB) procedure compared with the standard stapler (linear cutter) - separated mini-gastric bypass (LSSMGB). Additionally, surgical treatment will be compared with non-surgical treatment (hypocaloric diet therapy).

Who can participate? Obese adult patients with a BMI of between 30 kg/m2 and 50 kg/m2. What does the study involve? Participants are randomly allocated to one of three groups. Those in the first (A) group undergo the laparoscopic band-separated mini-gastric bypass procedure. Those in the second (B) group undergo the linear cutter stapler-separated mini-gastric bypass procedure. In three (C) group including standard lifestyle intervention on weight and hypocaloric diet therapy.

All patients are then followed up one month after surgery and again after 6 and, finally, 12 months after surgery where the changing body mass index, changes in co-morbidities, change telomere length and quality of life are assessed.

DETAILED DESCRIPTION:
Study hypothesis:

The increase in life expectancy depends on the degree of weight loss and the degree of regression of metabolic syndrome manifestations.

Ethics approval May 24, 2018, Ethics Committee of the Corporate Fund "University medical center".

Study design:

The interventional prospective randomized controlled clinical trial single-center study

Primary study design:

Interventional.

Secondary study design:

Randomised controlled trial.

Trial setting:

Hospitals.

Trial type:

Treatment.

Patient information sheet:

Not available in web format, please use contact details to request a participant information sheet.

Condition:

Morbid obesity.

Intervention type:

Procedure/Surgery

Background The prevalence of obesity in Kazakhstan in 2017 was more than 20% of the population. The annual increase in obesity rates over the past five years was 3.9 percent. Metabolic syndrome (MetS), which is based on abdominal adiposity, is a complex of symptoms that are risk factors for cardiovascular disease, manifestations of type 2 diabetes or prediabetes, non-alcoholic fatty liver disease, and dyslipidemia. Clinical MetS play a leading role in reducing the life expectancy and mortality of Kazakhstan's population.

Metabolic Surgery is the best option for treat type 2 diabetes and other components of MetS.

Reduction of excess body weight positively affects the clinical course and life expectancy of patients with MetS. Currently, surgeries and physicians accumulated positive results of treatment of patients with MetS methods of surgical and nonsurgical weight loss. The use of endoscopic staplers for surgical weight loss does not exclude the emergence of serious complications of surgery, for example, including bleeding and leakage in the stapler suture line. Therefore, the advantages of using a band in the gastric bypass surgery are justified from a security standpoint.

It is known that increased systemic inflammation and oxidative stress associated with obesity can accelerate aging and therefore telomere length (TL) can serve as an indicator of aging at the cellular level. Obesity has a known association with shorter TL. And weight loss in obese men is associated with increased telomere length. But the reduction in body weight with obesity changes the life expectancy remains not clear enough.

Study design The study is designed as an interventional, prospective, randomized, controlled, single-center clinical trial. Patient enrollment started on May 24, 2018, and the last patient is expected to be included in the study on September 4, 2019. The ethics committee of the Corporate Fund "University Medical Center" (UMC) has granted ethics approval for this study (May 24, 2018, Approval Number 5.

Study population/participants and recruitment Recruitment will be carried out by responsible bariatric surgeons with a minimum of 10 years of bariatric experience in the Department of Surgery, National Scientific Center for Oncology and Transplantation (Astana, Kazakhstan). Screening is done on the day - 7~ 0 prior to the treatment in order to ensure that patients fulfill the inclusion criteria. Patients will attend an informational meeting, where they will be informed about the study's purpose, process, and possible profits and risks. Patients fulfilling the study criteria who have signed the informed consent form will start treatment in accordance with the standard routines of the trial site. The informed consent will be obtained by the investigators. During the trial, the investigators will continue to provide additional health care or compensation for participants' health care needs that arise as a direct consequence of trial participation.

Randomization Informed consent will be obtained from each participant before patient enrollment in the study. Patients who meet all the inclusion criteria and none of the exclusion criteria will be consecutively included and randomized into one of the three study arms by the study statistician, who is not involved in the enrollment, assignment, or assessment of patients, on random allocation. Allocation concealment is ensured with the use of sequentially numbered, identical, opaque, sealed envelopes. The intervention will be assigned by a nurse, who has also no involvement in the enrollment or assessment of patients, who will open the sealed envelope during the visit before surgery.

* Group 1(A). The patients in Group 1 are treated by laparoscopic band-separated (stapleless) mini-gastric bypass procedure: Gastric band (absorbable ligature) introduced in the abdomen and retracted through the retro-gastric tunnel. Mobilization gastric fundus and creates obstructive gastroplication.
* Group 2(B). The patients in Group 2 are treated by Linear cutter stapler-separated mini-gastric bypass (MGB/OAGB): standard surgery.
* Group 3(C). The patients in Group 3 are treated by hypocaloric diet therapy with energy restriction (-500 kcal/d).

Blinding In this study, the single-party independent evaluation method is used to evaluate the outcomes of the study. The Outcome analyzer and the study statistician are in the masking state.

General procedure and monitoring Data collection and management Treatment-related data are collected at V1 (before intervention), at V2 (start of intervention). Follow-up data according to the study protocol will be followed from V1 to months 6 (V3) and 12 (V4). Data collection begins on the day a participant signs the informed consent and continues until the termination of the trial or until the participant withdraws from the trial at any time for any reason. If participants discontinue or deviate from the study protocols, the investigators will make best efforts to keep all missing data to a minimum. All original data are kept in chronological order for verification. Original data are timely transferred to a paper-based case report form (CRF) and an electronic database system located in a guarded facility at the trial site. Access to the study data is restricted. The PI will have access to the final dataset. All data files have a complete audit trail.

Statistical methods Sample size The sample size of this superiority trial was estimated based on the literature and our own unpublished data.

Data analysis Normally distributed variables will be expressed as their mean and standard deviation (SD) and non-normally distributed variables will be expressed as their median and interquartile range; categorical variables will be expressed as the sample size number plus a percentage (n, %). In test groups of continuous normally distributed variables, the Student t-test will be used; the Mann-Whitney U test will be used for continuous non-normally distributed data. Categorical variables will be compared with the χ2 test or Fisher's exact test or, when appropriate, as the relative risk. Statistical analysis will be conducted on an intention-to-treat (ITT) basis. The multivariable analysis will be conducted by logistic regression and a generalized mixed linear regression model to take into account any possible confounding covariate adjustments necessary, and also to consider within-center variability. A p-value of < 0.05 will be considered statistically significant.

Populations for evaluation and missing data management

All evaluations, in particular, the evaluation of the primary outcome measure, will be made on the basis of all randomized patients, regardless of whether or not they adhered to the treatment protocol or provided complete data sets. In particular, these latter patients are those:

Who discontinued the clinical trial; they will be evaluated as if they had complied with it Whose planned examinations were not carried out within the planned timeframe; they will still be taken into consideration in the analysis Patients who withdraw their consent to use their personal data for statistical analyses will be excluded from the analysis.

Missing reports of individual responses on the Quality-of-Life Questionnaire II will be replaced by simple imputation according to the recommendations of the test manual.

The reason for the missing data will be analyzed, and the data missing at random will be handled with multiple imputations and model-based approaches, such as mixed models or weighted generalized estimating equations (GEEs) for repeatedly measured outcomes. Sensitivity analysis will be performed to examine the robustness of the results to assumptions made in the complete case analysis.

Adverse events An adverse event (AE) refers to any untoward event that occurs during the clinical study but does not necessarily have a causal relationship with surgical treatment. Safety evaluation is carried out from the point at which the signature of the informed consent is obtained until the end of the study or until patient withdrawal from the trial, according to management requirements. Adverse events or serious adverse events should be reported.

A serious adverse event (SAE) refers to an event that causes hospitalization, prolonged hospitalization, disability, incapacity, life-threatening illness or death, or congenital malformation during the clinical trial.

During the study, all AEs are recorded. Records include the name of the AE (using standard medical terminology), the date of the AE occurrence, and disappearance/stability, severity, impact on the surgery, relationship with the surgery, treatment measures, and outcomes. If an SAE occurs, researchers fill in an SAE Report. The report is signed and dated and reported to the ethics committee of the Corporate Fund "University Medical Center" (UMC) and the clinical research center of the National Scientific Center for Oncology and Transplantation (Astana, Kazakhstan) within 24 h.

Quality control All surgeons and analyzers will be required to undergo special training prior to the trial to guarantee consistent practice. The training program will include diagnosis, inclusion/exclusion/exit criteria, surgery techniques, follow-up procedures, and completion of CRFs. The trial will be monitored by quality assurance personnel from the clinical research center of the National Scientific Center for Oncology and Transplantation, who will be independent of the study team, and an independent steering committee. There will be periodic monitoring to guarantee accuracy and quality throughout the study period. The essential documents (consent information, enrollment, protocol deviations, number and proportion of missed visits, and losses to follow-up) will be monitored and checked for accuracy and completeness by the monitors.

ELIGIBILITY:
Inclusion Criteria:

* BMI from 30 to 50 kg / m2;
* Metabolic syndrome (MetS) with abdominal adiposity if there are at least two components of MetS from the following: Increase in fasting plasma glucose: detected before diabetes (HbA1 = 5.7-6.4 or 3-fold increase in fasting plasma glucose:> 5.6 mmol / l); or previously diagnosed type 2 diabetes (HbA1> 6.5, or glucose> 6.1); Arterial hypertension AD 130 / 85 mmHg or receiving antihypertensive therapy; Increased triglyceride levels> 1.7 mmol / L or a specific treatment for this disorder; Reduction of high-density lipoproteins (HDL-C) <1.03 mmol / L in men and less than 1.29 mmol / L in women or receiving treatment for this disorder;
* The possibility of treatment for 12 months and the possibility of follow up;
* Informed written consent of the patient for randomization and treatment.

Exclusion Criteria:

* Age is less than 18 or more than 65 years;
* BMI less than 30 kg / m2 and more than 50 kg / m2;
* Drug addiction and alcohol consumption;
* Complete immobilization of the patient (paresis / paralysis);
* Presence in the anamnesis bariatric procedures;
* Insulin-dependent diabetes;
* Mental disorders or taking antidepressants;
* Socially vulnerable categories (according to ethical principles);
* Patients who do not understand the purpose of the study;
* Lack of informed written consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Change of body mass index | Baseline, at 12 months after surgery
  The measure is assessing a change of body mass index. Weight (kg) and height (cm) will be combined with the report of measurement by body mass index (BMI) kg/m2.

SECONDARY OUTCOMES:
Changes of comorbidities | Baseline, at 12 months after surgery
  Changes in co-morbidities by evaluation variable before and after intervention
Changes in the length of leukocyte telomere | Baseline, at 12 months after surgery
  To determine changes in the length of leukocyte telomer (TL) in patients of three groups
Change of Quality of life | at 12 months after surgery
  Quality of life, measured by the quality of life questionnaire the Moorehead-Ardelt Quality of Life Questionnaire II. 6 key areas were examined: self-esteem, physical well-being, social relationships, work, sexuality and eating behavior.The sum of these 6 scores generates an overall QoL score. Each score is classified into 5 categories (very poor: -3.0 to -2.1; poor: -2.0 to -1.1; fair: -1.0 to +1.0; good: 1.1 to 2.0: and very good: 2.1 to 3.0).the Quality of life of patients after weight loss is estimated as follows:
  * Poor ≤1
  * Satisfactory> 1 to 3
  * Good> 3 to 5
  * Very good > 5 to 7
  * Excellent> 7 to 9

CONTACTS AND LOCATIONS:
Overall Officials: Oral B Ospanov, Prof., Principal Investigator — Corporate fund "University Medical Center" (UMC)
Locations (1):
- National Scientific Center for Oncology and Transplantation, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ospanov OB. Laparoscopic Band-Separated One Anastomosis Gastric Bypass. Obes Surg. 2016 Sep;26(9):2268-2269. doi: 10.1007/s11695-016-2281-2. PMID 27384682
- [Derived] Ospanov O, Akilzhanova A, Buchwald JN, Fursov A, Bekmurzinova F, Rakhimova S, Yeleuov G, Kozhamkulov U, Abdina Z, Fursov R, Jumayeva L. Stapleless vs Stapled Gastric Bypass vs Hypocaloric Diet: a Three-Arm Randomized Controlled Trial of Body Mass Evolution with Secondary Outcomes for Telomere Length and Metabolic Syndrome Changes. Obes Surg. 2021 Jul;31(7):3165-3176. doi: 10.1007/s11695-021-05454-2. Epub 2021 May 8. PMID 33963974
- [Derived] Ospanov O, Yeleuov G, Kadyrova I, Bekmurzinova F. The life expectancy of patients with metabolic syndrome after weight loss: study protocol for a randomized clinical trial (LIFEXPE-RT). Trials. 2019 Apr 8;20(1):202. doi: 10.1186/s13063-019-3304-9. PMID 30961631